CLINICAL TRIAL: NCT04949048
Title: Evaluation of the Safety and Performance of Magneto PE Kit for Endovascular Thrombectomy in Patients With Acute Pulmonary Embolism
Brief Title: Evaluation of the Safety and Performance of Magneto PE Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magneto Thrombectomy Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT1-CLN001
Record Dates: First submitted 2021-01-03; First posted 2021-07-02 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magneto PE Kit (Experimental): Treatment with Magneto PE Kit
  Interventions: Device: Magneto PE Kit

INTERVENTIONS:
Device: Magneto PE Kit — All enrolled patients will be treated with Magneto PE Kit

SUMMARY:
This study is designed as a prospective, multi-center, multinational open labeled, single armed study to evaluate the safety and performance of the Magneto PE Kit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs, symptoms and presentation consistent with acute PE
* PE symptom duration ≤ 14 days
* CTA evidence of PE
* RV/LV ratio ≥ 0.9
* Heart rate <130 BPM prior to procedure
* Subject medically eligible for interventional procedure
* Age ≥ 18 and <75 years
* Consent process is completed

Exclusion Criteria:

* Thrombolytic use within 14 days
* Known bleeding diathesis or coagulation disorder
* Any contraindication to systemic therapeutic doses of heparin or other anticoagulants
* Hemodynamic collapse at presentation
* Decompensated heart failure
* Presence of Extra-Corporeal Membrane Oxygenation.
* Major trauma ISS> 15 within 14 days
* Cardiovascular or pulmonary surgery within last 7 days
* FiO2 requirement > 40% or > 6 LPM to keep oxygen saturation > 90%
* Hematocrit < 28%
* Platelets < 100,000/µL
* Serum creatinine > 1.8 mg/dL
* INR>2
* Left bundle branch block
* PAP > 70 mmHg m
* Imaging evidence suggests subject is not appropriate for mechanical thrombectomy
* Presence of intracardiac lead in right ventricle or atrium.
* Pacemaker or Implantable Cardioverter Defibrillator
* Presence of intracardiac thrombus
* Anaphylactic reaction to radiographic contrast agents that cannot be pre-treated
* Known right- to-left shunt,
* Known left ventricular ejection fraction ≤ 30%
* History of severe chronic pulmonary arterial hypertension
* History of underlying lung disease with oxygen dependence
* History of chest irradiation
* History of Heparin Induced Thrombocytopenia (HIT)
* Female who is pregnant or nursing
* Current participation in another investigational drug or device treatment study
* Life expectancy of < 90 days as determined by the investigator
* Subjects who are intubated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety of Magneto PE Kit | 48 (±8) hours
  Number of patients with a composite of major adverse events within 48 (± 8) hours of the index procedure

SECONDARY OUTCOMES:
Assessment of the safety of Magneto PE Kit | 30 (±3) days
  Number of patients with a composite of major adverse events within 30 (± 3) days of the index procedure
Assessment of ease of use during the procedure | Procedure
  Ease of use of Magneto PE Kit as assessed by a subjective questionnaire to be completed by the primary operator after the procedure
Assessment of the impact on RV dysfunction (RV/LV ratio) | 48 (±8) hours
  RV/LV ratio assessment at 48 (±8) hours

CONTACTS AND LOCATIONS:
Locations (5):
- Aarhus Univeristy Hospital, Aarhus, Denmark
- Israel (2):
  - Hadassah Ein Karem Hospital, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Poland (2):
  - John Paul II Hospital, Krakow
  - Poznan University Hospital, Poznan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen A, Musialek P, Araszkiewicz A, Schultz J, Nielsen-Kudsk JE, Tekieli L, Zajdel W, Slawek-Szmyt S, Taff Y, Weinberg I. First-in-Human Trial of Mechanical-Electric Thrombectomy in Acute Pulmonary Embolism. JACC Cardiovasc Interv. 2023 Mar 13;16(5):623-625. doi: 10.1016/j.jcin.2022.12.021. Epub 2023 Feb 8. No abstract available. PMID 36922052